CLINICAL TRIAL: NCT00402116
Title: Phase 1/2 Study of Enzastaurin Plus Temozolomide During and Following Radiation Therapy in Patients With Newly Diagnosed Glioblastoma Multiforme or Gliosarcoma
Brief Title: Phase 1/2 Study of Enzastaurin in Newly Diagnosed Glioblastoma Multiforme (GBM) and Gliosarcoma (GS) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9815; H6Q-MC-S008 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — enzastaurin; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): The Phase 1 consisted of the dose escalation of enzastaurin in 2 cohorts of up to 6 patients to assess maximum tolerated dose (MTD). Cohort 1 = radiotherapy/enzastaurin 250 mg per day/temozolomide 75 mg/m^2 therapy. The 6 initial cohort patients were clinically evaluated for dose-limiting toxicities (DLT). If no more than 1 of 6 patients experienced a DLT or tumor progression, patients continued 1 complete adjuvant enzastaurin/temozolomide 28-day cycle. If there was no significant toxicity after the first adjuvant cycle, participants received subsequent adjuvant enzastaurin/temozolomide cycles. If no more than 1 of the 6 initial cohort participants treated at 250 mg of enzastaurin experienced a DLT during radiotherapy and the first adjuvant cycle, up to 6 more participants could be entered at 500 mg of enzastaurin. The Phase 2, using the MTD determined in the Phase 1 (250 mg), evaluated the combination's safety and measured OS.
  Interventions: Drug: enzastaurin; Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: enzastaurin — Phase 1 - 250 mg Cohort 1 with one dose escalation allowed to 500 mg for Cohort 2, oral, daily, 6 weeks then twelve 28 day cycles
  Phase 2 - Phase 1 established dose, oral, daily, 6 weeks then twelve 28 day cycles
  Other Names: LY317615
Drug: temozolomide — 75 milligrams per meter squared (mg/m^2), oral, daily, 6 weeks then 200 mg/m^2, oral, daily, twelve 28 day cycles
Radiation: radiation therapy — 1.8-2.0 Gy x 30 fractions, 5 days/week, for 6 weeks

SUMMARY:
There will be 2 phases in this study. Patients will either be enrolled to the first phase or to the second phase, depending upon when they enroll into the study.

The first phase of this study is done to evaluate the safety of enzastaurin in patients. This is done by gradually increasing the dose of the drug in small groups of patients and watching closely for side effects.

In the second phase of the study, the dose determined to be safe will be used with temozolomide during and following radiation therapy to see if the combination can help patients with brain tumors live longer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of intracranial glioblastoma multiforme (GBM) or gliosarcoma (GS).
* Biopsy or resection must have been performed no more than 5 weeks prior to treatment.
* An MRI or CT scan must be obtained within 14 days prior to treatment.
* Patients must not have received prior drug therapy for brain tumors.
* Patients must have adequate organ function demonstrated by lab tests within 14 days prior to treatment.

Exclusion Criteria:

* Patients will be excluded if unable to swallow tablets.
* Patients will be excluded if unable to discontinue use of enzyme inducing antiepileptic drugs or have been off of these agents less than 2 weeks prior to treatment (i.e. phenytoin (Dilantin®), carbamazepine, etc.).
* Patients will be excluded if have active infection.
* Patients will be excluded if have a significant medical illness that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients will be excluded if they have concurrent therapy with an anticoagulant. If the patient requires anticoagulant therapy after starting treatment, the patient may remain on study but should be monitored carefully.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Francisco, California, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 participants entered Phase 1 of the study. A total of 60 participants were analyzed in Phase 2 for a total of 72 participants for both phases.
Groups:
- Phase 1- Cohort 1 (250 mg Enzastaurin): Phase 1--Determination of the maximum tolerated dose (MTD) of enzastaurin in participants with newly diagnosed GBM or GS receiving a 250 mg dose - Cohort 1.
- Phase 1 Cohort 2 (500 mg Enzastaurin): Phase 1--Determination of the maximum tolerated dose (MTD) of enzastaurin in participants with newly diagnosed GBM or GS receiving a 500 mg dose - Cohort 2.
- Phase 2: Phase 1 established dose (250 mg), daily for 6 weeks, then twelve 28-day cycles.
Period: Overall Study
Arm/Group | Phase 1- Cohort 1 (250 mg Enzastaurin) | Phase 1 Cohort 2 (500 mg Enzastaurin) | Phase 2
Started | 6 | 6 | 60
Completed | 3 | 0 | 5
Not Completed | 3 | 6 | 55
Not completed — Jaw infection after surgery-other | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 5
Not completed — Treatment completed per protocol | 1 | 1 | 2
Not completed — other complicating disease | 0 | 0 | 2
Not completed — Disease Progression | 0 | 4 | 38
Not completed — mistaken thrombocytopenia | 0 | 0 | 1
Not completed — decline related hyponatremia/tumor | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Phase 1- Cohort 1 (250 mg Enzastaurin): Participants who received 250 mg enzastaurin in Phase I with 75 mg/m^2 temozolomide and radiotherapy.
- Phase 1 Cohort 2 (500 mg Enzastaurin ): Participants who received 500 mg enzastaurin in Phase I with 75 mg/m^2 temozolomide and radiotherapy.
- Phase 2: Participants who received 250 mg enzastaurin in Phase II with 75 mg/m^2 temozolomide and radiotherapy.
- Total: Total of all reporting groups
Arm/Group | Phase 1- Cohort 1 (250 mg Enzastaurin) | Phase 1 Cohort 2 (500 mg Enzastaurin ) | Phase 2 | Total
Number analyzed (Participants) | 6 | 6 | 60 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (7.54) | 52.5 (13.84) | 55.3 (10.95) | 54.7 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 17 | 21
  Male | 5 | 3 | 43 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 4 | 5
  White | 6 | 3 | 52 | 61
  Unknown | 0 | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 60 | 72

OUTCOME MEASURES:

1. Primary Outcome: Phase 1- Determination of the Maximum Tolerated Dose (MTD) of Enzastaurin
Description: Phase 1- dose escalation of enzastaurin in 2 cohorts up to 6 participants each in order to assess MTD. After radiation/enzastaurin 250 mg per day/temozolomide 75 mg/m^2 therapy, if no more than 1 of 6 patients experienced a dose-limiting toxicity (DLT) or tumor progression, participants completed one 28-day cycle. If no significant toxicity after the first cycle, participants received subsequent cycles. If no more than 1 of the 6 patients treated at 250 mg of enzastaurin experienced a DLT, up to 6 more patients could be entered at escalated dose cohort of enzastaurin (500 mg).
Time Frame: Until MTD can be determined (up to 12 cycles, 28 days per cycle)
Population: All Phase I participants who received at least one dose of study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- Phase 1 Participants: Participants who received escalating doses of 250 mg and 500 mg enzastaurin in Phase 1 with 75 mg/m^2 temozolomide and radiotherapy.
Arm/Group | Phase 1 Participants
Number analyzed (Participants) | 12
milligrams (mg) | 250

2. Primary Outcome: Phase 1 and Phase 2 - Overall Survival (OS)
Description: OS is the time from surgical diagnosis to the date of death from any cause. For participants who were alive, OS was censored at the last contact.
Time Frame: Baseline to death from any cause (Up to 48 weeks)
Population: Phase 2 participants combined with Phase 1 cohort 1 participants who also received 250 mg enzastaurin.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- 250 mg Enzastaurin Phases 1 and 2 Combined: Phase 2 participants combined with Phase 1 - Cohort 1 participants who also received 250 mg enzastaurin.
Arm/Group | 250 mg Enzastaurin Phases 1 and 2 Combined
Number analyzed (Participants) | 66
months | 18.3 [15.2 to 19.3]

3. Secondary Outcome: Phase 1 - Number of Participants With Adverse Events (AEs)
Description: Summaries of serious AEs (SAEs) and all other non-serious AEs are located in the Reported Adverse Event Module.
Time Frame: Every cycle (up to 12 cycles, 28 days per cycle)
Population: All Phase I participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1- Cohort 1 (250 mg Enzastaurin): Summaries of SAEs and all other non-serious AEs for Phase 1- Cohort 1 (250 mg Enzastaurin) participants
- Phase 1 Cohort 2 (500 mg Enzastaurin ): Summaries of SAEs and all other non-serious AEs for Phase 1- Cohort 2 (500 mg Enzastaurin) participants
Arm/Group | Phase 1- Cohort 1 (250 mg Enzastaurin) | Phase 1 Cohort 2 (500 mg Enzastaurin )
Number analyzed (Participants) | 6 | 6
Participants | 0 | 1

4. Secondary Outcome: Phase 1 and 2: Association Between Biomarkers and Clinical Outcome
Description: Phosphorylated-S6 (pS6) ribosomal protein is a biomarker that's being investigated as a potential marker for clinical outcome using 2211 or 2215 antibody to pS6. Reported here are the hazard ratios and 95% confidence intervals (CIs) for participants for whom an pS6 immunohistochemistry (IHC) score was available. The IHC assays were scored using a 0 to +3 scoring system (no positive staining was scored 0; at least 25% immunoreactivity of cells was scored +1; 26% to 75% was scored +2; and 76% or greater was scored +3). Hazard ratio (HR) > 1 indicates worse outcome for that IHC score.
Time Frame: Baseline, Cycle 2, end of study (up to 12 cycles, 28 days per cycle)
Population: Combined Phases 1 and 2 populations for whom IHC scores were obtained. HR > 1 indicates poorer overall survival for that IHC score.
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Groups:
- 250 mg Enzastaurin Phases 1 and 2 Combined: Participants with valid IHC scores from combined Phase 1 and 2 populations 250 mg enzastaurin.
Arm/Group | 250 mg Enzastaurin Phases 1 and 2 Combined
Number analyzed (Participants) | 49
Hazard ratio
  S6 2211 score | 1.70 [1.05 to 2.77]
  S6 2215 score | 1.69 [1.08 to 2.66]

5. Secondary Outcome: Phase 1 - Response Rate With Macdonald Criteria
Description: Response categories: complete response (CR): disappearance of all enhancing tumor on consecutive magnetic resonance imaging (MRI) scans at least 1 month apart, off steroids, and neurologically stable or improved. Partial response (PR): 50% reduction in size of enhancing tumor on consecutive MRI scans at least 1 month apart, steroids stable or reduced, and neurologically stable or improved. Progressive disease (PD): >25% increase in size of enhancing tumor or any new tumor on MRI scans, or neurologically worse, and steroids stable or increased. Stable disease (SD): all other situations.
Time Frame: Baseline, following radiation, every other cycle (up to 12 cycles, 28 days per cycle)
Population: Efficacy analysis in phase I was not conducted. Instead, participants who took 250mg in phase I were pooled with phase II participants and are presented in other outcome measures (2 and 8, respectively) in this record. Thus there were 0 participants for this measure.
Groups:
- 250 mg Enzastaurin Phases 1 and 2 Combined: Efficacy analysis in Phase 1 was not conducted. Instead, participants who took 250 mg enzastaurin in Phase 1 were pooled with Phase 2 participants. Overall survival (OS) and progression-free survival (PFS) for this combined group are presented in other outcome measures (2 and 8, respectively) in this result record.
Arm/Group | 250 mg Enzastaurin Phases 1 and 2 Combined
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 2 - Number of Participants With Adverse Events (AEs)
Description: Summaries of serious AEs (SAEs) and all other non-serious AEs are located in the Reported Adverse Event Module.
Time Frame: Every cycle (28 days per cycle)
Population: All Phase 2 participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 - 250 mg Enzastaurin: Summaries of SAEs and all other non-serious AEs for Phase 2 - 250 mg Enzastaurin participants are located in the Reported Adverse Event Module.
Arm/Group | Phase 2 - 250 mg Enzastaurin
Number analyzed (Participants) | 60
Participants | 22

7. Secondary Outcome: Number of Participants Undergoing Magnetic Resonance Imaging/Magnetic Resonance Spectroscopy (MRI/MRS) for Clinical Evaluation at Baseline
Description: Number of patients having MRI/MRS for clinical evaluation with baseline assessment.
Time Frame: Each radiologic assessment (up to 12 cycles, 28 days per cycle)
Population: 35 patients underwent MRI and had baseline measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 - 250 mg: Participants who underwent magnetic resonance imaging (MRI) for clinical evaluation and had a baseline assessment.
Arm/Group | Phase 2 - 250 mg
Number analyzed (Participants) | 35
Participants | 35

8. Secondary Outcome: Phase 1 and 2 - Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of first dose to the first observation of disease progression, or death due to any cause.
Time Frame: Baseline to measured progressive disease (up to 12 cycles, 28 days per cycle)
Population: Phase 2 participants combined with Phase 1 cohort 1 participants who also received 250 mg enzastaurin.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- 250 mg Enzastaurin Phases 1 and 2 Combined: All treated participants in the 250 mg enzastaurin cohort from Phases 1 and 2 combined
Arm/Group | 250 mg Enzastaurin Phases 1 and 2 Combined
Number analyzed (Participants) | 66
months | 10.6 [8.4 to 12.7]

9. Secondary Outcome: Functional Assessment of Cancer Therapy - Brain (FACT-Br)
Description: Total FACT-Br score includes physical well-being, social/family well-being, emotional well-being, functional well-being and additional concerns related to brain tumors. The score ranges 0 to 200, with a higher score representing better quality of life.
Time Frame: Every cycle (up to 12 cycles, 28 days per cycle)
Population: All treated participants who received at least one dose of study drug in the 250 mg enzastaurin cohort from Phases 1 and 2 combined and who also provided FACT-Br data from at least 1 visit (N = 65). One participant lacked these data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 250 mg Enzastaurin Phases 1 and 2 Combined
Number analyzed (Participants) | 65
units on a scale
  Baseline visit | 153.5 (24.08)
  Radiation therapy visit | 156.1 (23.30)
  Cycle 1 | 151.9 (26.87)
  Cycle 2 | 152.0 (30.67)
  Cycle 3 | 158.9 (22.10)
  Cycle 4 | 158.8 (24.48)
  Cycle 5 | 158.3 (26.30)
  Cycle 6 | 159.0 (26.46)
  Cycle 7 | 164.1 (19.45)
  Cycle 8 | 163.6 (23.19)
  Cycle 9 | 162.0 (21.89)
  Cycle 10 | 159.3 (27.02)
  Cycle 11 | 158.2 (24.98)
  Cycle 12 | 163.5 (26.67)

10. Secondary Outcome: M.D. Anderson Symptom Inventory - Brain Tumor (MDASI-BT)
Description: General and brain tumor-specific symptoms each assessed on a scale of 0 to 10, with a higher score representing higher symptom burden. The 4 symptom scales reported as changing over the course of the study are listed here.
Time Frame: Every cycle (up to 12 cycles, 28 days per cycle)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enzastaurin 250 mg Phases 1 and 2 Combined-Fatigue: All treated participants who received at least 1 dose of study drug in the 250 mg enzastaurin cohort from Phases 1 and 2 combined and provided MDASI-BT data from at least 1 visit. Question: Your fatigue (tiredness) at its WORST?
- Enzastaurin 250 mg Phase 1 and 2 Combined-Memory: All treated participants who received at least 1 dose of study drug in the 250 mg enzastaurin cohort from Phases 1 and 2 combined and provided MDASI-BT data from at least 1 visit (N = 65). Question: Your problem with remembering things at its WORST?
- Enzastaurin 250 mg Phase 1 and 2 Combined-Appetite: All treated participants who received at least 1 dose of study drug in the 250 mg enzastaurin cohort from Phases 1 and 2 combined and provided MDASI-BT data from at least 1 visit. Question: Your problem with lack of appetite at its WORST?
- Enzastaurin 250 mg Phase 1 and 2 Combined-Concentration: All treated participants who received at least 1 dose of study drug in the 250 mg enzastaurin cohort from Phases 1 and 2 combined and provided MDASI-BT data from at least 1 visit. Question: Your difficulty concentrating at its WORST?
Arm/Group | Enzastaurin 250 mg Phases 1 and 2 Combined-Fatigue | Enzastaurin 250 mg Phase 1 and 2 Combined-Memory | Enzastaurin 250 mg Phase 1 and 2 Combined-Appetite | Enzastaurin 250 mg Phase 1 and 2 Combined-Concentration
Number analyzed (Participants) | 65 | 65 | 65 | 65
units on a scale
  Baseline | 2.4 (2.1) | 1.8 (2.6) | 0.3 (1.1) | 1.2 (1.9)
  Radiation therapy visit | 3.3 (2.1) | 2.2 (2.3) | 1.0 (1.9) | 1.4 (1.7)
  Cycle 1 | 3.6 (2.5) | 2.4 (2.6) | 1.6 (2.4) | 1.8 (2.2)
  Cycle 2 | 3.7 (2.7) | 2.5 (3.0) | 1.8 (2.5) | 1.9 (2.2)
  Cycle 3 | 3.2 (2.5) | 2.0 (1.9) | 1.4 (2.3) | 1.5 (1.8)
  Cycle 4 | 2.6 (2.1) | 1.9 (1.6) | 1.0 (1.8) | 1.5 (1.6)
  Cycle 5 | 3.3 (2.5) | 2.1 (2.4) | 0.6 (1.6) | 1.6 (2.1)
  Cycle 6 | 2.9 (2.4) | 1.6 (1.3) | 0.7 (1.2) | 1.2 (1.7)
  Cycle 7 | 2.8 (2.4) | 1.4 (1.3) | 0.7 (1.4) | 1.3 (1.6)
  Cycle 8 | 2.6 (2.4) | 1.4 (1.5) | 0.5 (0.9) | 1.1 (1.3)
  Cycle 9 | 2.8 (2.5) | 1.8 (1.6) | 1.0 (1.9) | 1.1 (1.5)
  Cycle 10 | 1.9 (1.9) | 1.5 (1.9) | 0.4 (1.2) | 1.2 (1.3)
  Cycle 11 | 3.0 (2.8) | 1.6 (2.6) | 0.2 (0.6) | 0.9 (1.6)
  Cycle 12 | 1.7 (1.8) | 1.2 (0.9) | 0.4 (0.7) | 1.2 (1.6)

11. Secondary Outcome: Phase 1- Pharmacokinetics (PK): Maximum Observed Drug Concentration During 1 Dosing Interval at Steady State (Cmax,ss) for Enzastaurin, LY326020, and Total Analyte (Enzastaurin + LY326020) When Enzastaurin Administered With or Without Temozolomide
Description: Cmax,ss was calculated using concentration versus time data of enzastaurin, LY326020, and Total Analyte (enzastaurin + LY326020) when 250 mg or 500 mg enzastaurin was administered alone or with 75 mg/m^2 temozolomide. Data are reported as Geometric Mean and Geometric Coefficient of Variation (%).
Time Frame: Cycle 1 Day 22, Cycle 2 Day 5, 28 days per Cycle
Population: Pharmacokinetic analyses were conducted for individual participants who received at least one dose of study drug and had pharmacokinetic samples collected. One participant dose was reduced from 500 mg to 250 mg after Cycle 1 Day 1 so is included in the 250 mg dose group (N=7).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole per liter (nmol/L)
Groups:
- Enzastaurin 250 mg: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 1 Day 22 (enzastaurin alone) following enzastaurin 250 mg oral (po) daily QD) for Phase 1 Cohort 1.
- Enzastaurin 250 mg + Temozolomide: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 2 Day 5 (enzastaurin with temozolomide) following enzastaurin 250 mg oral (po) daily QD) for Phase 1 Cohort 1.
- Enzastaurin 500 mg: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 2 Day 5 (enzastaurin alone) following enzastaurin 500 mg oral (po) daily QD) for Phase 1 Cohort 2.
- Enzastaurin 500 mg + Temozolomide: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 2 Day 5 (enzastaurin with temozolomide) following enzastaurin 500 mg oral (po) daily QD) for Phase 1 Cohort 2.
Arm/Group | Enzastaurin 250 mg | Enzastaurin 250 mg + Temozolomide | Enzastaurin 500 mg | Enzastaurin 500 mg + Temozolomide
Number analyzed (Participants) | 7 | 6 | 3 | 3
nanomole per liter (nmol/L)
  Enzastaurin | 504 (52) | 458 (41) | 1350 (149) | 719 (114)
  LY326020 | 370 (38) | 392 (27) | 198 (274) | 465 (87)
  Total Analyte | 853 (44) | 821 (28) | 1570 (159) | 1010 (114)

12. Secondary Outcome: Phase 1 and 2- Pharmacokinetics: Area Under the Concentration-Time Curve During 1 Dosing Interval at Steady State (AUCτ,ss) for Enzastaurin, LY326020 and Total Analyte (Enzastaurin + LY326020) When Enzastaurin Administered With or Without Temozolomide
Description: AUCτ,ss was calculated using concentration versus time data of enzastaurin, LY326020, and total analyte (enzastaurin + LY326020). Data are reported as Geometric Mean and Geometric Coefficient of Variation (%).
Time Frame: Phase 1, Cycle 1 Day 22, Cycle 2 Day 5 of a 28 day Cycle; Phase 2, Cycle 1 Day 22 of a 28 day Cycle
Population: Pharmacokinetic analyses were conducted for individual participants who received at least one dose of study drug and had pharmacokinetic samples collected. In Phase I, one participant dose was reduced from 500 mg to 250 mg after Cycle 1 Day 1 so was included in 250 mg dose group (N=7).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol•h/L
Groups:
- Enzastaurin 250 mg Phase 1: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 1 Day 22 (enzastaurin alone) following enzastaurin 250 mg orally (po) daily (QID) for Phase 1 Cohort 1.
- Enzastaurin 250 mg + Temozolomide: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 2 Day 5 (enzastaurin with temozolomide) following enzastaurin 250 mg po QID for Phase 1 Cohort 1.
- Enzastaurin 250 mg Phase 2: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 1 Day 22 (enzastaurin alone) following enzastaurin 500 mg oral po QID for Phase 1 Cohort 2
- Enzastaurin 500 mg: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 2 Day 5 (enzastaurin with temozolomide) following enzastaurin 500 mg oral po QID for Phase 1 Cohort 2.
- Enzastaurin 500 mg + Temozolomide: Enzastaurin, LY326020 and total analyte (enzastaurin + LY326020) on Cycle 1 Day 22 (enzastaurin alone) following enzastaurin 250 mg oral po QID for Phase 2.
Arm/Group | Enzastaurin 250 mg Phase 1 | Enzastaurin 250 mg + Temozolomide | Enzastaurin 250 mg Phase 2 | Enzastaurin 500 mg | Enzastaurin 500 mg + Temozolomide
Number analyzed (Participants) | 7 | 6 | 33 | 3 | 3
nmol•h/L
  Enzastaurin | 5390 (57) | 5270 (36) | 7720 (91) | 16600 (274) | 10100 (133)
  LY326020 | 7260 (35) | 7380 (22) | 12800 (38) | 4240 (283) | 8650 (95)
  Total Analyte | 12800 (41) | 12800 (19) | 21400 (53) | 21300 (256) | 18900 (114)

ADVERSE EVENTS:
Groups:
- Phase 1- Cohort 1 (250 mg Enzastaurin): Phase 1--Determination of the maximum tolerated dose (MTD) of enzastaurin in participants with newly diagnosed GBM or GS receiving a 250 mg dose.
- Phase 1 Cohort 2 (500 mg Enzastaurin): Phase 1--Determination of the maximum tolerated dose (MTD) of enzastaurin in participants with newly diagnosed GBM or GS receiving a 500 mg dose.
- Phase 2 - 250 mg Enzastaurin: Participants received 250 mg enzastaurin daily for 6 weeks, then twelve 28-day cycles.
Arm/Group | Phase 1- Cohort 1 (250 mg Enzastaurin) | Phase 1 Cohort 2 (500 mg Enzastaurin) | Phase 2 - 250 mg Enzastaurin
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 22/60
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1- Cohort 1 (250 mg Enzastaurin) (N=6) | Phase 1 Cohort 2 (500 mg Enzastaurin) (N=6) | Phase 2 - 250 mg Enzastaurin (N=60)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic leakage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Complex partial seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myelitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1- Cohort 1 (250 mg Enzastaurin) (N=6) | Phase 1 Cohort 2 (500 mg Enzastaurin) (N=6) | Phase 2 - 250 mg Enzastaurin (N=60)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 16 (16)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) | 52 (52)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Auditory disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 5 (5)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 3 (3)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (4) | 42 (42)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5)
Feces discolored (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 34 (34)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 14 (14)
Calcinosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Edema (General disorders) | 0 (0) | 0 (0) | 3 (3)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 5 (5)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 6 (6) | 52 (52)
Fever (General disorders) | 2 (2) | 0 (0) | 2 (2)
Flu-like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 13 (14)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1) | 4 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 5 (5)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 9 (9)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 14 (14)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 10 (10)
Creatinine increased (Investigations) | 2 (2) | 2 (2) | 6 (6)
Ear, nose and throat examination abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin (Investigations) | 3 (3) | 1 (1) | 29 (29)
Hemoglobin decreased (Investigations) | 2 (2) | 3 (3) | 13 (13)
International normalized ratio (Investigations) | 1 (1) | 0 (0) | 2 (2)
Leukocyte count decreased (Investigations) | 2 (2) | 1 (1) | 30 (30)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (3) | 7 (7)
Neutrophils (Investigations) | 1 (1) | 0 (0) | 11 (11)
Platelet count decreased (Investigations) | 5 (5) | 3 (3) | 12 (12)
Platelets decreased (Investigations) | 2 (2) | 3 (3) | 23 (23)
Proctoscopy abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 3 (3) | 0 (0) | 3 (3)
Weight loss (Investigations) | 2 (2) | 3 (3) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 26 (26)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 38 (39)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 6 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 9 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 12 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 13 (13)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 8 (8)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 13 (13)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 6 (6)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 13 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 3 (3) | 5 (5)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 7 (7)
Convulsion (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 7 (7)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 29 (29)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 4 (4) | 2 (2) | 20 (20)
Neurologic disorder NOS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 11 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 3 (3) | 9 (9)
Speech disorder (Nervous system disorders) | 1 (1) | 2 (2) | 11 (11)
Taste alteration (Nervous system disorders) | 3 (3) | 0 (0) | 12 (12)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 6 (6)
Visual field defect (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 11 (11)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 10 (10)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 14 (14)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 20 (20)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 5 (5)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 4 (4) | 4 (4) | 8 (8)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 41 (41)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 8 (8)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Vascular disorder (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days